CLINICAL TRIAL: NCT04141995
Title: A Phase IIa (Pilot) Study of Neoadjuvant Chemotherapy With Folinic Acid, 5-FU, Irinotecan and Oxaliplatin (FOLFIRINOX) With Digoxin in Patients With Resectable Pancreatic Cancer
Brief Title: FOLFIRINOX With Digoxin in Patients With Resectable Pancreatic Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to low accrual and futility
Sponsor: University of Nebraska (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0668-19-FB; 1P50CA127297-01A2 (NIH)
Record Dates: First submitted 2019-10-18; First posted 2019-10-28 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-04

CONDITIONS: Pancreas Cancer; Adenocarcinoma of the Pancreas
Keywords: Resectable
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Digoxin; Fluorouracil; Leucovorin; Irinotecan; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Treatment (Experimental): Participants start FOLFIRINOX. They will also begin digoxin and take it up to 4-5 months time period in patients with resectable pancreatic cancer. Digoxin is taken at the time of neo-adjuvant chemotherapy treatment, prior to surgery. After surgery, participants will continue with post-adjuvant chemotherapy.
  Interventions: Drug: Digoxin; Drug: 5Fluorouracil; Drug: Calcium Leucovorin; Drug: Irinotecan; Drug: Oxaliplatin

INTERVENTIONS:
Drug: Digoxin — Tablet, Oral: Generic: 0.125 mg, 0.25 mg
  Other Names: Lanoxin; Digitek; Digox
Drug: 5Fluorouracil — 5-FU will be given as a 46 hour continuous IV infusion
  Other Names: Adrucil; 5-FU
Drug: Calcium Leucovorin — IV injection over 90 minutes
  Other Names: Folinic Acid
Drug: Irinotecan — IV administration over 90 minutes
  Other Names: Camptothecin-11; CPT-11; Camptosar
Drug: Oxaliplatin — IV administration
  Other Names: Eloxatin

SUMMARY:
The purpose of this study is to determine the feasibility and safety of combining digoxin as a modulator of the hypoxia pathway in combination with FOLinic acid, 5-Fluorouracil, IRINotecan and OXaliplatin (FOLFIRINOX) in participants with resectable pancreatic cancer.

DETAILED DESCRIPTION:
Participants with resectable pancreatic cancer will be treated with oxaliplatin 85 mg/m² IV over 2 hours, irinotecan 150 mg/m² given concurrently with folinic acid 400 mg/m² IV over 90 min, followed by a 46-hour infusion of 5-fluorouracil 2400 mg/m². Slow oral digitalization will be used starting with a daily dose of 0.125 (participants over age 65) or 0.25 mg (participants 65 or younger) per mouth daily. A steady-state will be achieved after five half-lives, which is about 7 to 10 days in the average participant. The initial blood level will be obtained one week after starting digoxin. Assuming the digoxin level is at steady-state and the renal function is stable, there is a linear relationship between digoxin dose and serum concentration. The target digoxin level is between 0.8 to 1.2 ng/mL. Participants will receive IV chemotherapy at 2 week intervals. Re-staging imaging will be performed after 4 doses. If the participants has stable or responsive disease, an additional 4 doses will be given followed by re-staging imaging. The participant will then undergo surgical exploration ~ 4 weeks after the last dose of chemotherapy.

The primary endpoint is clinical toxicity. Other endpoints are status of pathologic margins, response rate, pathologic stage, progression-free survival, and overall survival. The correlative endpoint is baseline exome sequencing of circulating cell free tumor DNA. Measurement of quantity of circulating cell free tumor DNA at 4 week intervals while on chemotherapy and prior to surgery; resume at 3 month intervals after surgery. Genomic DNA will be collected at baseline for pharmacogenetic studies of polymorphisms that may be pertinent for the drugs used in the study. Blood will be collected for analysis of possible biomarkers of response to digoxin modulation.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed pancreatic adenocarcinoma. Participants must have resectable disease with no evidence of distant metastasis.
* 19 years of age or older.
* Eastern Cooperative Oncology Group (ECOG) Performance Scale (PS) of 0-1 (fully active to restricted in strenuous activity).
* Chemotherapy for malignancies other than pancreatic cancer completed > 5 years ago and is no evidence of the prior malignancy at time of study entry.
* Radiographically assessable disease.
* Initial absolute neutrophil count (ANC) greater than or equal to 1000/μL and platelet count greater than or equal to 100,000/μL.
* Normal serum potassium, magnesium and corrected calcium level.
* Serum creatinine less than or equal to 2.0 mg/dL.
* Total bilirubin <= 1.5 mg/dL [unless the participant has Gilbert disease with elevated non-conjugated (indirect) bilirubin; in such cases, the indirect bilirubin should be <= 1.0 mg/dL].
* If participant has biliary obstruction, biliary decompression will be required. Either endoscopic placement of biliary stent or percutaneous transhepatic drainage are acceptable. Once biliary drainage has been established, institution of FOLFOX therapy may proceed when the total bilirubin falls to <= 5.0 mg/dL. The addition of irinotecan will be delayed until the total bilirubin is 1.5 mg/dL or lower.
* Awareness of the neoplastic nature of his/her disease and willingly provide written, informed consent after being informed of the procedure to be followed, the experimental nature of the therapy, alternatives, potential benefits, side-effects, risks, and discomforts.
* No prior chemotherapy for pancreatic cancer.

Exclusion Criteria:

* Unable to undergo staging laparoscopy, such as a prior history of multiple abdominal operations in which laparoscopy may not be technically feasible or might be potentially harmful.
* A contra-indication to receiving digoxin therapy (e.g., AV block, sick sinus syndrome, bradycardia, hypersensitivity to digoxin or digitalis preparations).
* Uncontrolled inter-current illness including, but not limited to ongoing or active infection requiring intravenous antibiotics, symptomatic congestive heart failure, unstable angina pectoris, or serious, uncontrolled cardiac arrhythmia, that might jeopardize the ability of the participant to receive the therapy in this study with reasonable safety.
* Pregnant and nursing women (risk posed by chemotherapy agents). Female participants of childbearing potential must have a negative urine pregnancy test before receiving the first dose of study drug.
* Prior malignancy except for adequately treated basal cell or squamous cell skin cancer, adequately treated non-invasive carcinomas, or other cancers from which the participant has been disease-free least 5 years.
* Known HIV infection or active hepatitis B or C infection (concern for increased toxicity).
* Active autoimmune disease [e.g., rheumatoid arthritis (RA), systemic lupus erythematosus (SLE), ulcerative colitis (UC), Crohn's Disease, multiple sclerosis (MS), ankylosing spondylitis (AS)].
* Recognized acquired, hereditary, or congenital immunodeficiency disease including cellular immunodeficienciess, hypogammaglobulinemia, or dysgammaglobulinemia.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2021-02-12 (Actual); Primary Completion 2025-05-13 (Actual); Study Completion 2025-05-13 (Actual)

PRIMARY OUTCOMES:
Number of patients able to undergo resection surgery | 16 weeks
  Regimen will be considered for further investigation if 14 of the 20 patients are able to undergo resection

SECONDARY OUTCOMES:
Percentage of subjects with grade 4 thrombocytopenia and grade 3-4 diarrhea | 16 weeks
  Continuous monitoring will be performed to monitor toxicity using Pocock stopping boundary that yields the probability of crossing the boundary at most 0.05 when the toxicity rate is equal to 0.182 or 0.28 separately.

CONTACTS AND LOCATIONS:
Overall Officials: Jean Grem, MD, Principal Investigator — University of Nebraska
Locations (1):
- University of Nebraska Medical Center, Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No